CLINICAL TRIAL: NCT04732325
Title: CRCNS: Model-based Characterization of Spinal Cord Stimulation for Pain
Brief Title: Sensory Testing of Multiple Forms of Spinal Cord Stimulation for Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Scott Lempka, Associate Professor, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: HUM00164430; R01AT010817 (NIH)
Record Dates: First submitted 2021-01-27; First posted 2021-02-01 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Chronic Pain; Failed Back Surgery Syndrome; Complex Regional Pain Syndromes; Neuropathic Pain
Keywords: Spinal cord stimulation
MeSH Terms: conditions — Chronic Pain; Failed Back Surgery Syndrome; Complex Regional Pain Syndromes; Neuralgia | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Intervention Model Description: Subjects will receive each treatment for seven days following one of six randomly-allocated sequences
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: There will be two research teams. One team will be unblinded (e.g., clinical care provider/company representative, study coordinator) and will perform stimulator programming/adjustment, and the other team will be blinded (e.g., research personnel) and will perform clinical testing and collect study outcome measures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (6):
- Burst / kHz / Sham / Tonic (Experimental): Participants will be randomized to one of six treatment arms. Participants will receive burst, kHz, tonic, and sham spinal cord stimulation (SCS). Each treatment will be applied for a duration of seven days. Participants will be blinded during programming.
  Interventions: Device: Spinal cord stimulation
- Burst / Sham / kHz / Tonic (Experimental): Participants will be randomized to one of six treatment arms. Participants will receive burst, kHz, tonic, and sham spinal cord stimulation (SCS). Each treatment will be applied for a duration of seven days. Participants will be blinded during programming.
  Interventions: Device: Spinal cord stimulation
- kHz / Sham / Burst / Tonic (Experimental): Participants will be randomized to one of six treatment arms. Participants will receive burst, kHz, tonic, and sham spinal cord stimulation (SCS). Each treatment will be applied for a duration of seven days. Participants will be blinded during programming.
  Interventions: Device: Spinal cord stimulation
- kHz / Burst / Sham / Tonic (Experimental): Participants will be randomized to one of six treatment arms. Participants will receive burst, kHz, tonic, and sham spinal cord stimulation (SCS). Each treatment will be applied for a duration of seven days. Participants will be blinded during programming.
  Interventions: Device: Spinal cord stimulation
- Sham / Burst / kHz / Tonic (Experimental): Participants will be randomized to one of six treatment arms. Participants will receive burst, kHz, tonic, and sham spinal cord stimulation (SCS). Each treatment will be applied for a duration of seven days. Participants will be blinded during programming.
  Interventions: Device: Spinal cord stimulation
- Sham / kHz / Burst / Tonic (Experimental): Participants will be randomized to one of six treatment arms. Participants will receive burst, kHz, tonic, and sham spinal cord stimulation (SCS). Each treatment will be applied for a duration of seven days. Participants will be blinded during programming.
  Interventions: Device: Spinal cord stimulation

INTERVENTIONS:
Device: Spinal cord stimulation — Researchers will program the spinal cord stimulation (SCS) system to deliver, according to the randomization status of the participant, burst, kHz, tonic, and sham stimulation.

SUMMARY:
Doctors sometimes treat chronic pain with devices that send mild electrical currents into the spinal cord. This type of treatment is referred to as neurostimulation. A common form of neurostimulation therapy is spinal cord stimulation (SCS). In this study, researchers want to learn more about how SCS affects pain processing and relieves pain. The researchers will examine multiple forms of SCS in chronic pain patients who are receiving SCS from their own doctors as part of their standard of care. During the study, participants will be asked to complete a variety of evaluations at certain time points.

ELIGIBILITY:
Inclusion criteria:

* Chronic intractable pain of the trunk and/or limbs
* Undergoing SCS as part of standard clinical care for chronic pain management
* Candidates will have been implanted with a commercial SCS device
* Candidates who are 18 years or older and can speak, read, and understand English
* Able to understand study procedures and to comply with them for the entire length of the study
* Must be willing to participate in COVID-19 symptom screening and answer questions about COVID-19 diagnosis 1-3 days before a scheduled visit
* Must be willing to wear a face-covering during all study visits

Exclusion criteria:

* Subjects who are pregnant or nursing
* Subjects with current, habitual, or previous use within the last 12 months of artificial nails, nail enhancements, or nail extensions that cover any portion of either thumbnail
* Subjects who are unable or unwilling to cooperate with clinical testing
* Subjects having any impairment, activity or situation that in the judgment of study personnel would prevent satisfactory completion of the study protocol
* Inability or unwillingness of individual or legal guardian/representative to give written informed consent
* Subjects who currently have or tested positive in the last 14 days for COVID-19, or are symptomatic for COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-09-11 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
SCS-induced changes in temporal summation (TS) | Baseline (At randomization) and at the end of each seven-day treatment
  TS refers to an increased perception of pain in response to sequential stimuli of equal physical strength. At the end of each treatment period, TS scores will be calculated by subtracting the average pain rating of the single-stimulus trials from the average pain rating of the ten-stimuli trials. If the difference is a positive number, the researchers will conclude that there was pain summation, where larger numbers will indicate increased pain summation or TS. If the difference is zero or a negative number, the researchers will conclude that there was no pain summation or TS.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Lempka, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to share IPD at this time.

DOCUMENTS (1):
  • Informed Consent Form (2023-06-11): https://cdn.clinicaltrials.gov/large-docs/25/NCT04732325/ICF_000.pdf